CLINICAL TRIAL: NCT02216539
Title: Interest of Learning Self-hypnosis for Patients Awaiting Lung Transplantation
Acronym: AUTOHYPNOSE-TP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change of sponsor
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014-A00538-39
Record Dates: First submitted 2014-08-13; First posted 2014-08-15 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Lung Diseases
Keywords: All terminal; leading; indication; lung transplantation
MeSH Terms: conditions — Lung Diseases | interventions — Hypnosis; Lung Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Self-hypnosis (Experimental): Patients trained to self-hypnosis before surgery
  Interventions: Behavioral: Self-hypnosis; Procedure: Lung transplantation; Other: Standard post-operative pain management
- Usual pain management (Active Comparator): Patients receiving the usual post-operative pain management protocols
  Interventions: Procedure: Lung transplantation; Other: Standard post-operative pain management

INTERVENTIONS:
Behavioral: Self-hypnosis — Patients will be trained to self-hypnosis prior to surgery, in order to be able to use self-hypnosis as a pain-management tool after surgery
  Arms: Self-hypnosis
Procedure: Lung transplantation
Other: Standard post-operative pain management — Post-operative pain management treatments as per usual protocols in the hospital

SUMMARY:
Patients benefitting from a lung transplantation are subject to long-lasting and often severe post-operative pain. Self-hypnosis has been proven effective in the management of acute pain.

The study hypothesis is that pre-operative training in self-hypnosis given to patients awaiting lung transplantation, will result in a reduction of post-operative pain one month after surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients over 15 years of age
* indication of lung transplantation

Exclusion Criteria:

* patient unable to receive training in self-hypnosis (for cognitive, linguistic or cultural reasons)

Ages: 15 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Average Pain Score (Visual Analog Scale) One Month After Surgery | one month after transplantation
  Average level of pain (scored by the patient on a visual analog scale), during the 48 hours preceding the scheduled consultation at one month post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mireille Michel-Cherqui, MD, Principal Investigator — Hôpital Foch, Suresnes, France; Marc Fischler, MD, Study Chair — Hôpital Foch, Suresnes, France
Locations (1):
- Hôpital Foch, Suresnes, France